CLINICAL TRIAL: NCT01862406
Title: The Impact of Generic Labels on Consumption Dosage and Medication Compliance
Brief Title: The Impact of Generic Labels on Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Marco Aurelio Bianchini, Associate Professor of Dentistry, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UFSC-CEPSH-649-322600
Record Dates: First submitted 2013-05-16; First posted 2013-05-24 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Generic Label; Brand-name Label
MeSH Terms: interventions — Drug Labeling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic Label (Experimental): Purportedly generic version of the analgesic presented
  Interventions: Other: Label
- Brand-name Label (Active Comparator): actual brand-name analgesic presented
  Interventions: Other: Label

INTERVENTIONS:
Other: Label — Participants were presented with either a generic label or a brand-name label

SUMMARY:
Although generic drugs are pharmacologically equivalent to their brand-name counterparts, prejudices against the former remain strong among patients and doctors. In a randomized controlled field experiment, this research assesses the extent to which generic (versus brand-name) labels affect patients' consumption dosage, medication compliance and reported pain.

DETAILED DESCRIPTION:
One hundred one patients scheduled to undergo invasive dental surgeries (i.e., dental implants) participated in the experiment. After dental surgery, patients were prescribed a once-daily analgesic regimen for up to 7 days. The intervention consisted of label manipulation. Patients were randomly assigned to either the brand-name analgesic or to its (purportedly) cheaper generic version. In reality, all participants obtained the same brand-name medication. The medication was provided at no cost, and patients were instructed to take the first pill while at the clinic. They were informed that they could (a) increase the dosage of the prescribed analgesic to twice daily if necessary and (b) stop taking the medication when no longer needed. Any other changes to the regimen were discouraged, and patients were instructed to consult with the dentist before any such changes. Telephone follow-ups were conducted at 24 hours, 4 days, and 7 days after surgery. Two main dependent variables were obtained: the number of prescribed analgesics consumed and the number of non-prescribed analgesics consumed. The patients also reported the pain felt during the period.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo dental implants and/or bone graft surgeries at the UFSC dental clinic

Exclusion Criteria:

* Patients not scheduled to undergo these treatments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Non-Compliance | 1 day after the intervention
  Number of patients who consumed at least one non-prescribed analgesic pill during the first 24 hours
Non-Compliance | 4 days after the intervention
  Number of patients who consumed at least one non-prescribed analgesic pill during the period (from day 2 to day 4)
Non-compliance | 7 days after the intervention
  Number of patients who consumed at least one non-prescribed analgesic pill during the period (from day 5 to day 7)

SECONDARY OUTCOMES:
Consumption Dosage | 1 day after the intervention
  Average number of pills consumed during the study period (first 24 hours)
Consumption Dosage | 4 days after the intervention
  Average number of pills consumed during the study period (from day 2 to day 4)
Consumption dosage | 7 days after the intervention
  Average number of pills consumed during the study period (from day 5 to 7)

OTHER OUTCOMES:
Pain levels | 1 day after the intervention
  Average retrospective and current level of pain; eleven-point scale (0=not at all, 10=extreme)
Pain levels | 4 days after the intervention
  Average retrospective and current level of pain; eleven-point scale (0=not at all, 10=extreme)
Pain levels | 7 days after the intervention
  Average retrospective and current level of pain; eleven-point scale (0=not at all, 10=extreme)
Perceived Efficacy | 1 day after the intervention
  perceived efficacy of prescribed painkiller (0=It does not reduce pain at all; 10=it eliminates pain completely)
Perceived Efficacy | 4 days after the intervention
  perceived efficacy of prescribed painkiller (0=It does not reduce pain at all; 10=it eliminates pain completely)
Perceived Efficacy | 7 days after the intervention
  perceived efficacy of prescribed painkiller (0=It does not reduce pain at all; 10=it eliminates pain completely)
Referral | 1 day after the intervention
  the likelihood of indicating it a friend (0=Never; 10=Certainly).
referral | 4 days after the intervention
  the likelihood of indicating it a friend (0=Never; 10=Certainly).
referral | 7 days after the intervention
  the likelihood of indicating it a friend (0=Never; 10=Certainly).